CLINICAL TRIAL: NCT05227664
Title: A Phase II Study of AK117/AK112 in Combination With Chemotherapy for Patients With Previously Untreated Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of AK117/AK112 in Metastatic Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK117-203
Record Dates: First submitted 2022-01-27; First posted 2022-02-07 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Metastatic Triple-negative Breast Cancer; Locally Advanced Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Taxes; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cohort1(AK117 +AK112 +Nab-Paclitaxel/ Paclitaxel) (Experimental): Subjects receive AK117 and AK112 Plus Nab-Paclitaxel/ Paclitaxel until disease progression or unacceptable toxicity.
  Interventions: Drug: AK117; Drug: AK112; Drug: Nab paclitaxel; Drug: paclitaxel
- cohort2(AK117 +Nab-Paclitaxel/ Paclitaxel) (Experimental): Subjects receive AK117 Plus Nab-Paclitaxel/ Paclitaxel until disease progression or unacceptable toxicity.
  Interventions: Drug: AK117; Drug: Nab paclitaxel; Drug: paclitaxel
- cohort3(AK112 +Nab-Paclitaxel/ Paclitaxel) (Experimental): Subjects receive AK112 Plus Nab-Paclitaxel/ Paclitaxel until disease progression or unacceptable toxicity.
  Interventions: Drug: AK112; Drug: Nab paclitaxel; Drug: paclitaxel

INTERVENTIONS:
Drug: AK117 — Intravenous (IV) infusion
  Arms: cohort1(AK117 +AK112 +Nab-Paclitaxel/ Paclitaxel); cohort2(AK117 +Nab-Paclitaxel/ Paclitaxel)
Drug: AK112 — Intravenous (IV) infusion
  Arms: cohort1(AK117 +AK112 +Nab-Paclitaxel/ Paclitaxel); cohort3(AK112 +Nab-Paclitaxel/ Paclitaxel)
Drug: Nab paclitaxel — Nab-Paclitaxel at a starting dose of 100 milligrams per square meter via IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.
Drug: paclitaxel — Paclitaxel at a starting dose of 90 milligrams per square meter via IV infusion on Days 1, 8, and 15 of each 28-day cycle until disease progression or unacceptable toxicity.

SUMMARY:
This trial is a Phase II study. The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of AK117/AK112 administered with chemotherapy in participants with locally advanced or metastatic triple-negative breast cancer (TNBC) who have not received prior systemic therapy for metastatic breast cancer (mBC).

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced, histologically documented TNBC characterized by absence of human epidermal growth factor 2 (HER2), estrogen receptor (ER), and progesterone receptor (PR) expression
* No prior chemotherapy or targeted systemic therapy for inoperable locally advanced or metastatic TNBC
* Eligible for taxane monotherapy
* A representative formalin-fixed, paraffin-embedded tumor specimen in paraffin blocks, or at least 5 unstained slides with an associated pathology report documenting ER, PR, and HER2 negativity.
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Measurable disease as defined by RECIST v1.1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Known central nervous system (CNS) disease, except for asymptomatic CNS metastases
* Leptomeningeal disease
* Pregnancy or lactation
* History of autoimmune disease
* Prior allogeneic stem cell or solid organ transplantation
* Positive test for human immunodeficiency virus
* Active hepatitis B or hepatitis C
* Receipt of a live, attenuated vaccine within 30 days prior to randomization, during treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , based on RECIST v1.1
Number of participants with adverse events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Up to approximately 2 years
  Disease control rate (DCR) is defined as the proportion of subjects with CR, PR, or stable disease(SD) based on RECIST V1.1
Duration of response (DOR) | Up to approximately 2 years
  DOR is defined for participants who had an objective response as the time from the first occurrence of a documented unconfirmed response (CR or PR) to the date of disease progression per RECIST v1.1 or death from any cause, whichever occurred first
Time to response (TTR) | Up to approximately 2 years
  TTR is defined for participants who had an objective response as the time from the start of treatment to the first occurrence of a documented unconfirmed response (CR or PR) .
Progression-free survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the start of treatment till the first documentation of disease progression (per RECIST v1.1 criteria) assessed by the investigator or death due to any cause (whichever occurs first).
Overall survival (OS) | Up to approximately 2 years
  Overall survival is defined as the time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Hunan Cancer Hospital, Changsha
  - Xiangyang Central Hospital, Xiangyang